CLINICAL TRIAL: NCT05548049
Title: A Prospective Randomized Trial Comparing Conventional And Piezosurgery Method In Mandibular Bone Block Harvesting From The Retromolar Region
Brief Title: Autogenous Ramus Bone Block Harvesting With Piezosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assistant Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUDHF_FB_002
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Alveolar Bone Resorption
MeSH Terms: interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery Group (Experimental): In the experimental group, a piezosurgical device was used to harvest the bone block from the ramus area.
  Interventions: Device: Bone harvesting from ramus area with piezosurgery for autogenous bone augmentation
- Conventional Group (Active Comparator): In the experimental group, a conventional burr was used to harvest the bone block from the ramus area.
  Interventions: Device: Bone harvesting from ramus area with conventional burs for autogenous bone augmentation

INTERVENTIONS:
Device: Bone harvesting from ramus area with piezosurgery for autogenous bone augmentation — In this invervention, the piezo-surgical device settings were set to irrigation: '4', function: 'cortical', light: 'auto'. After the full-thickness flap was lifted with the periosteal elevator, superior and vertical osteotomies were performed with the OT-12 piezo-surgical tip. Lower horizontal osteotomies were performed using OT8-L or OT-8-R piezo tips according to the studied quadrant, combining the vertical osteotomy.
  Arms: Piezosurgery Group
Device: Bone harvesting from ramus area with conventional burs for autogenous bone augmentation — In control group, After the full-thickness flap is lifted with the periosteal elevator, using a thin #9 fissure burand the surgical handpiece S-11 Straight tip , the physiodispenser settings are according to the manufacturer's recommendations. The osteotomy was performed after it was adjusted to 40,000 rpm as appropriate. Bone incisions were completed with a round bur to combine the lower horizontal osteotomies and 2 vertical osteotomies. The osteotomies were completed with the help of a thin flat drill, and the block graft was carefully separated from the donor site.
  Arms: Conventional Group

SUMMARY:
The aim of this randomized prospective clinical trial was to evaluate the outcome of bone block harvesting from the retromolar region using the Conventional and Piezosurgery Method.

The study was planned on 19 patients (13F,6M) on 31 donor sites. In patients with bilateral bone harvesting, the donor site and the surgical method to be used were determined by the randomization protocol, while in patients with bone harvesting from a single site, the donor site was determined by considering parameters such as proximity to the operation site and distance to the inferior alveolar nerve. Clinical parameters such as operation time, pain, swelling, trismus, nerve damage were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* The main inclusion criteria were severe alveolar ridge atrophy in the horizontal plane (≤4 mm) and no accompanying vertical defect, according to preoperative CBCT scans.

Exclusion Criteria:

* Individuals who had systemic disease affecting bone or soft tissue metabolism
* Smokers (more than 10 cigarettes a day
* Alcohol dependent
* Systemic disease affecting bone or soft tissue metabolism
* Donor field in the mouth of another region (simfiz, tuber etc.) or any extra-oral field is planned to be used
* Patients with cleft lip-palate or defect exceeding the alveolar crest
* Grafts applied to defects caused by tumors, osteoradionecrosis, or congenital malformations
* Patients with an unstable systemic condition such as metabolic bone disease, uncontrolled diabetes, or untreated hypothyroidism, as well as smokers, patients undergoing radiation therapy or chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Osteotomy time | Intraoperative
  The time from the start of the osteotomy to the luxation of the bone block was measured with the help of a digital stopwatch.

SECONDARY OUTCOMES:
Change in pain | 7 days
  Postoperative pain was assessed using a Visual Analogue Scale (VAS) ranging from the absence of pain (score 0) to the most severe pain imaginable
Change in Mouth opening | 7 days
  The distance between the mesio-incisal corners of the upper and lower central incisors was measured with the help of a ruler when the mouth opening was at its maximum.
Change in Oral Health-related Quality of Life | 14 days
  Evaluated by OHIP-14
Operation time | Intraoperative
  The total time from the first incision of the operation site to the last suture was measured with the help of a digital stopwatch as the operation time.
Change in facial swelling | 7 days
  With the technique described by Neupert ; Angle of mandible-tragus Angle of mandible-lateral canthus of eye Mandible corner-nose wing Angle of mandible oral-commissures Measurements were made with a tape measure from 5 points, with the mandible corner-pogonion.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available in 1 month and will be available for 2 years

REFERENCES:
- [Background] Silva FM, Cortez AL, Moreira RW, Mazzonetto R. Complications of intraoral donor site for bone grafting prior to implant placement. Implant Dent. 2006 Dec;15(4):420-6. doi: 10.1097/01.id.0000246225.51298.67. PMID 17172961
- [Background] Sohn DS, Ahn MR, Lee WH, Yeo DS, Lim SY. Piezoelectric osteotomy for intraoral harvesting of bone blocks. Int J Periodontics Restorative Dent. 2007 Apr;27(2):127-31. PMID 17514884
- [Background] Robiony M, Polini F, Costa F, Zerman N, Politi M. Ultrasonic bone cutting for surgically assisted rapid maxillary expansion (SARME) under local anaesthesia. Int J Oral Maxillofac Surg. 2007 Mar;36(3):267-9. doi: 10.1016/j.ijom.2006.08.013. Epub 2006 Nov 16. PMID 17112705
- [Background] Hanser T, Doliveux R. MicroSaw and Piezosurgery in Harvesting Mandibular Bone Blocks from the Retromolar Region: A Randomized Split-Mouth Prospective Clinical Trial. Int J Oral Maxillofac Implants. 2018 Mar/Apr;33(2):365-372. doi: 10.11607/jomi.4416. PMID 29534125
- [Background] Sittitavornwong S, Gutta R. Bone graft harvesting from regional sites. Oral Maxillofac Surg Clin North Am. 2010 Aug;22(3):317-30, v-vi. doi: 10.1016/j.coms.2010.04.006. PMID 20713265
- [Background] Pereira RS, Pavelski MD, Griza GL, Boos FBJD, Hochuli-Vieira E. Prospective evaluation of morbidity in patients who underwent autogenous bone-graft harvesting from the mandibular symphysis and retromolar regions. Clin Implant Dent Relat Res. 2019 Aug;21(4):753-757. doi: 10.1111/cid.12789. Epub 2019 May 16. PMID 31094060
- [Background] Chiapasco M, Casentini P, Zaniboni M. Bone augmentation procedures in implant dentistry. Int J Oral Maxillofac Implants. 2009;24 Suppl:237-59. PMID 19885448
- [Background] Starch-Jensen T, Deluiz D, Deb S, Bruun NH, Tinoco EMB. Harvesting of Autogenous Bone Graft from the Ascending Mandibular Ramus Compared with the Chin Region: a Systematic Review and Meta-Analysis Focusing on Complications and Donor Site Morbidity. J Oral Maxillofac Res. 2020 Nov 30;11(3):e1. doi: 10.5037/jomr.2020.11301. eCollection 2020 Jul-Sep. PMID 33262880
- [Background] Nkenke E, Neukam FW. Autogenous bone harvesting and grafting in advanced jaw resorption: morbidity, resorption and implant survival. Eur J Oral Implantol. 2014 Summer;7 Suppl 2:S203-17. PMID 24977256
- [Background] Nielsen HB, Starch-Jensen T. Lateral ridge augmentation in the posterior part of the mandible with an autogenous bone block graft harvested from the ascending mandibular ramus. A 10-year retrospective study. J Stomatol Oral Maxillofac Surg. 2021 Apr;122(2):141-146. doi: 10.1016/j.jormas.2020.05.020. Epub 2020 May 29. PMID 32480048
- [Background] Nkenke E, Stelzle F. Clinical outcomes of sinus floor augmentation for implant placement using autogenous bone or bone substitutes: a systematic review. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:124-33. doi: 10.1111/j.1600-0501.2009.01776.x. PMID 19663959
- [Derived] Bayram F, Demirci A. A randomized controlled trial comparing conventional and piezosurgery methods in mandibular bone block harvesting from the retromolar region. BMC Oral Health. 2023 Dec 9;23(1):986. doi: 10.1186/s12903-023-03739-9. PMID 38071300